CLINICAL TRIAL: NCT06299111
Title: A Master Protocol for a Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of REGN9933 and REGN7508, Monoclonal Antibodies Against Factor XI for Prevention of Venous Thromboembolism in Patients With a Peripherally Inserted Central Catheter (ROXI-CATH)
Brief Title: A Trial to Learn How Well REGN9933 and REGN7508 Work for Preventing Blood Clots, and How Safe They Are, in Adults Who Have a Peripherally Inserted Central Catheter (PICC)
Acronym: ROXI-CATH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R9933-DVT-2308; 2023-508603-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism
Keywords: Anti-factor XI (FXI) monoclonal antibody; Venous Thromboembolism; Peripherally inserted central catheter
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REGN9933 (Experimental): Randomized 1:1:1
  Interventions: Drug: REGN9933
- REGN7508 (Experimental): Randomized 1:1:1
  Interventions: Drug: REGN7508
- Placebo (Placebo Comparator): Randomized 1:1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN9933 — Intravenous (IV) single dose administered
  Arms: REGN9933
Drug: REGN7508 — IV single dose administered
  Arms: REGN7508
Drug: Placebo — IV single dose administered
  Arms: Placebo

SUMMARY:
This study is researching 2 different experimental drugs called REGN9933 and REGN7508 (called "study drugs"). The study is focused on adults undergoing a placement of a catheter in the vein, also called a 'PICC line'.

The aim of the study is to see how effective the study drug is at preventing venous thromboembolism (VTE) and other related disease after catheter placement.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. PICC is clinically indicated for at least 14 days and is anticipated to remain in place for at least 14 days
2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2 or equivalent functional status as described in the protocol
3. Body weight ≥45 kg and ≤130 kg during the screening period
4. International normalized ratio (INR) and aPTT values at or below the upper limit of normal as defined by the local lab during the screening period
5. Platelet count ≥100 x 10^9/L during the screening period as described in the protocol

Key Exclusion Criteria:

1. Unsuccessful PICC placement or any other complication associated with this procedure that in the opinion of the study investigator may present any safety concerns to the participant
2. History of prior venous thrombosis in the arm in which the PICC is to be placed
3. Peripheral catheter(s) in the same arm in which the PICC is to be placed or expected need for peripheral catheter(s) placement in the same arm the PICC is to be placed as described in the protocol
4. History of known thromboembolic disease or thrombophilia
5. Participants requiring therapeutic anticoagulation and/or antiplatelet therapy as described in the protocol
6. Expected to receive cancer therapy or other medication associated with a prior episode of Grade 4 thrombocytopenia as described in the protocol
7. Any history of intracranial or intraocular bleeding, excessive operative or post-operative bleeding, traumatic spinal or epidural anesthesia, or history of bleeding diathesis (such as but not limited to Hemophilia A or B, von Willebrand's disease, fibrinogen deficiency, and other inherited or acquired bleeding disorders) as described in the protocol

Note: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of confirmed VTE per central reading center (CRC) review | Through Day 14
Incidence of treatment-emergent adverse event (TEAEs) | Up to Day 100
Severity of TEAEs | Up to Day 100

SECONDARY OUTCOMES:
Incidence of confirmed PICC associated venous thrombosis per CRC review | Through Day 14
Incidence of major bleeding | Through Day 14
Incidence of clinically relevant non-major (CRNM) bleeding | Through Day 14
Concentrations of REGN9933 in serum | Up to Day 75
Concentrations of REGN7508 in serum | Up to Day 75
Change in activated partial thromboplastin time (aPTT) | Up to Day 75
Change in prothrombin time (PT) | Up to Day 75
Incidence of anti-drug antibody (ADA) to REGN9933 over time | Up to Day 75
Magnitude of ADA to REGN9933 over time | Up to Day 75
Incidence of ADA to REGN7508 over time | Up to Day 75
Magnitude of ADA to REGN7508 over time | Up to Day 75

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (23):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
- Sveta Sofia Hospital, Sofia, Bulgaria
- Canada (4):
  - Juravinski Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - University Health Network, Toronto, Ontario
- Israel (7):
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Soroka University Medical Center, Beersheba, Southern District
  - Hadassah University Medical Center, Jerusalem
  - Lanadio Medical Center, Netanya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Romania (2):
  - Arensia Research Clinic, Bucharest
  - Arensia Exploratory Medicine Clinic at Country Hospital Cluj-Napoca, Cluj-Napoca
- United Kingdom (3):
  - University hospital Southampton, Southampton, Hampshire
  - Cardiff and Vale University Health Board - University Hospital Wales, Cardiff, Wales
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: ROXI-CATH — https://roxicath.com/